CLINICAL TRIAL: NCT02526082
Title: Long-term Follow-up of the Helsinki Businessmen Study Cohort of Men Born in 1919-1934
Brief Title: Long-term Follow-up of the Helsinki Businessmen Study
Acronym: HBS
Status: Active, not recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Timo Strandberg, Professor, Helsinki University Central Hospital
Other Study IDs: HBS Group
Record Dates: First submitted 2015-06-10; First posted 2015-08-18 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Quality of Life; Syndromes; Aging; Cardiovascular Disease; Death
Keywords: cardiovascular disease; frailty; quality of life; mortality; prevention
MeSH Terms: conditions — Syndrome; Cardiovascular Diseases; Death; Frailty | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — APOE, telomeres, DNA collected for future use
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Total, observational: Various cardiovascular risk groups described below
- High-risk intervention: Healthy but at high risk in 1974
  Interventions: Other: Intervention
- High-risk control: Healthy but at high risk in 1974
- Low-risk conrtol: Healthy and at low risk in 1974
- Sick control: Medications or clinical disease in 1974
- Refused: Refused or no response in 1974

INTERVENTIONS:
Other: Intervention — Multifactorial intervention with lifestyle changes and drugs as needed
  Groups: High-risk intervention

SUMMARY:
The Helsinki Businessmen Study (HBS) is a clinico-epidemiological longitudinal study started in 1964. It also included a 5-year randomized, controlled multifactorial primary prevention trial of cardiovascular diseases between 1974-1980. The cohort is being actively followed-up through national registers since the 1980, and since 2000 with regular questionnaire surveys. Latest in 2015. Also clinical and laboratory studies have been performed in random subcohorts. Follow-up is ongoing with new hypothesis-generating research questions.

DETAILED DESCRIPTION:
The Helsinki Businessmen Study (HBS) was originally a convenient cohort of male executives and businessmen (born 1919-1934, n=3490), who participated in health check-ups between 1964-1973, but since the beginning of 1970s it has developed into a clinico-epidemiological longitudinal study. Primary focus was on the prevention of cardiovascular diseases (CVD), but since 2000 focus has been shifting to geriatrics, and with its long follow-up (up to 50 years) HBS can be seen as a "life-course" study. Traditional CVD risk factors are available from the 1960s and in 1974 participants (available n=3310) were divided in groups according to their clinical status and CVD risk. Two high-risk groups (n=1222) and low-risk group (n=593) participated in a 5-year multifactorial primary prevention study in 1974-1980 (in-trial and post-trial results have been published in 1985 and 1991). The whole original cohort has been followed-up from national registers since 1985 and with regular questionnaire surveys since 2000. Random subcohorts have been studied clinically with laboratory and genetic examinations in 2003 and 2011. The latest questionnaire survey was performed in winter 2015 by which two thirds of the original cohort had died. Follow-up of the cohort is ongoing and new research questions formulated..

ELIGIBILITY:
Inclusion Criteria:

* Participants of director studies at the Institute of Occupational Health in Helsinki, Finland, between 1964-1973

Exclusion Criteria:

* Non-participants

Ages: 31 Years to 46 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Originally a convenient cohort of male executives and businessmen (born 1919-1934, n=3490), who participated in health check-ups during 1964-1973, but since the beginning of 1970s it has developed into a clinic-epidemiological longitudinal study.
Sampling Method: Non-Probability Sample
Enrollment: 3490 (Actual)
Dates: Start 1964-01; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Total mortality: national registers | change from baseline up to 612 months

SECONDARY OUTCOMES:
Health-related quality of life: questionnaire data | change from baseline up to 612 months
Geriatric syndromes and disability: questionnaires, clinical examinations, registers | change from baseline up to 612 months
Morbidity: self-report, national registers, hospital and autopsy records | change from baseline up to 612 months
Medications: self-report, national registers | change from baseline up to 612 months
Cause-specific mortality: national registers, autopsy records | change from baseline up to 612 months

CONTACTS AND LOCATIONS:
Overall Officials: Timo E Strandberg, MD, Principal Investigator — Helsinki University Central Hospital

REFERENCES:
- [Result] Strandberg TE, Salomaa VV, Naukkarinen VA, Vanhanen HT, Sarna SJ, Miettinen TA. Long-term mortality after 5-year multifactorial primary prevention of cardiovascular diseases in middle-aged men. JAMA. 1991 Sep 4;266(9):1225-9. PMID 1870247
- [Result] Miettinen TA, Huttunen JK, Naukkarinen V, Strandberg T, Mattila S, Kumlin T, Sarna S. Multifactorial primary prevention of cardiovascular diseases in middle-aged men. Risk factor changes, incidence, and mortality. JAMA. 1985 Oct 18;254(15):2097-102. PMID 4046137
- [Result] Strandberg AY, Strandberg TE, Stenholm S, Salomaa VV, Pitkala KH, Tilvis RS. Low midlife blood pressure, survival, comorbidity, and health-related quality of life in old age: the Helsinki Businessmen Study. J Hypertens. 2014 Sep;32(9):1797-804. doi: 10.1097/HJH.0000000000000265. PMID 25014505
- [Derived] Strandberg TE, Pitkala KH, Kivimaki M. Sleep duration in midlife and old age and risk of mortality over a 48-year follow-up: The Helsinki businessmen study (HBS) cohort. Maturitas. 2024 Jun;184:107964. doi: 10.1016/j.maturitas.2024.107964. Epub 2024 Mar 8. PMID 38471293
- [Derived] Jyvakorpi SK, Urtamo A, Kivimaki M, Salomaa V, Strandberg TE. Association of midlife body composition with old-age health-related quality of life, mortality, and reaching 90 years of age: a 32-year follow-up of a male cohort. Am J Clin Nutr. 2020 Nov 11;112(5):1287-1294. doi: 10.1093/ajcn/nqaa230. PMID 32844221
- [Derived] Jyvakorpi SK, Urtamo A, Kivimaki M, Strandberg TE. Associations of protein source, distribution and healthy dietary pattern with appendicular lean mass in oldest-old men: the Helsinki Businessmen Study (HBS). Eur Geriatr Med. 2020 Aug;11(4):699-704. doi: 10.1007/s41999-020-00330-1. Epub 2020 May 22. PMID 32444996